CLINICAL TRIAL: NCT03782987
Title: Relative Bioavailability of a Single Oral Dose of BI 730357 When Administered Alone or in Combination With Multiple Oral Doses of Itraconazole in Healthy Male Subjects (an Open-label, One-way Crossover Study)
Brief Title: A Study in Healthy Men to Test How Itraconazole Influences the Amount of BI 730357 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1407-0014; 2018-003495-13 (EudraCT Number)
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Results first posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2022-08

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 730357 + Itraconazole (T) (Experimental): Participants were administered 50 mg BI 730357 tablet orally on Day 1 along with 20 mL of 10 mg/ mL Itraconazole oral solution in treatment period 2 only (T). Itraconazole was administered once daily for 12 days from Day -3 to Day 9.
  Interventions: Drug: BI 730357; Drug: Itraconazole
- BI 730357 (R) (Experimental): Participants were administered 50 mg BI 730357 tablet orally on Day 1 alone in treatment period 1 (R).
  Interventions: Drug: BI 730357

INTERVENTIONS:
Drug: BI 730357 — 0 mg BI 730357 tablet orally on Day 1
Drug: Itraconazole — 20 mL of 10 mg/ mL Itraconazole oral solution in treatment period 2 only (T). Itraconazole was administered once daily for 12 days from Day -3 to Day 9.
  Arms: BI 730357 + Itraconazole (T)

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of BI 730357 in plasma when given as oral single dose together with multiple oral doses of itraconazole (Test, T) as compared to when given alone as oral single dose (Reference, R)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant Electrocardiogram (ECG) finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

* Liver enzyme (ALT, AST, GGT) values above upper limit of normal at the screening examination
* History of drug-induced liver injury
* History of heart failure, or any evidence of ventricular dysfunction in the history
* History of hereditary fructose intolerance
* Male subjects with WOCBP partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of first administration of trial medication until 30 days after the last administration of trial medication
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, two-treatment, two-period, one-way crossover trial in healthy participants in order to compare the test treatment (T) to the reference treatment (R). All participants underwent treatment R in Period 1 (Visit 2) and treatment T in Period 2 (Visit 3). There was at least 10 days washout between the administrations of BI 730357.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist site which would then ensured that all participants met all inclusion/exclusion criteria. Participants were not to be entered to trial if any one of the specific entry criteria were not met.
Groups:
- BI 730357 Alone/ BI 730357+Itraconazole: Participants were administered 50 milligram (mg) BI 730357 tablet orally on Day 1 alone in treatment period 1 (R) and along with 20 milliliter (mL) of 10 mg/ mL Itraconazole oral solution on Day 1 of treatment period 2 (T). Itraconazole was administered once daily on Day -3, -2, -1 and 1 before administration of BI 730357 and on Day 2 to 9 in treatment period 2 only. There was a washout interval of at least 10 days between the administrations of BI 730357.
Period: Period 1
Arm/Group | BI 730357 Alone/ BI 730357+Itraconazole
Started (Started are treated) | 14
Completed | 14
Not Completed | 0
Period: Washout Period
Arm/Group | BI 730357 Alone/ BI 730357+Itraconazole
Started | 14
Completed | 14
Not Completed | 0
Period: Period 2
Arm/Group | BI 730357 Alone/ BI 730357+Itraconazole
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who received at least 1 dose of trial medication.
Arm/Group | BI 730357 Alone/ BI 730357+Itraconazole
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the BI 730357 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC0-tz, area under the concentration-time curve of the BI 730357 in plasma over the time interval from 0 to the last quantifiable data point is presented.
Time Frame: Pharmacokinetic samples were taken within 3 hours (h) before administration of BI 730357 and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 34, 47, 71, 119 and 167 h in both periods and additionally at 215 and 263 h only for period 2.
Population: Pharmacokinetic (PK) parameter set (PKS): The PKS included all subjects of the TS who provided at least 1 primary or secondary PK parameter that was not excluded due to relevant protocol deviations or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: Nanomole* hour/ Litre (nmol*h/ L)
Arm/Group | BI 730357 + Itraconazole (T) | BI 730357 (R)
Number analyzed (Participants) | 14 | 14
Nanomole* hour/ Litre (nmol*h/ L) | 43239.08 (NA) — Standard Error is Geometric standard error (gSE) = 1.09 | 6657.49 (NA) — Standard Error is Geometric standard error (gSE) = 1.09
Statistical Analysis 1: Comparison: BI 730357 + Itraconazole (T) vs BI 730357 (R); Statistical model was an analysis of variance (ANOVA) on the logarithmic scale including 'subjects' as random effect and 'treatment' as fixed effect; Test type: Other; Geometric mean (gMean) ratio (%) (T/ R) = 649.48, 90% CI 2-sided [541.29 to 779.29], Standard Error of Mean 27.7 — Confidence intervals were calculated based on the residual error from the ANOVA. Standard error of the mean is actually intra-individual geometric coefficient of variance (gCV)

2. Primary Outcome: Maximum Measured Concentration of the BI 730357 in Plasma (Cmax)
Description: Cmax, maximum measured concentration of the BI 730357 in plasma is presented here.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol/ L
Arm/Group | BI 730357 + Itraconazole (T) | BI 730357 (R)
Number analyzed (Participants) | 14 | 14
nmol/ L | 311.01 (NA) — Standard Error is Geometric standard error (gSE) = 1.07 | 186.36 (NA) — Standard Error is Geometric standard error (gSE) = 1.07
Statistical Analysis 1: Comparison: BI 730357 + Itraconazole (T) vs BI 730357 (R); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean ratio (%) (T/ R) = 166.88, 90% CI 2-sided [148.42 to 187.64], Standard Error of Mean 17.7 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Area Under the Concentration-time Curve of the BI 730357 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞, area under the concentration-time curve of the BI 730357 in plasma over the time interval from 0 extrapolated to infinity is presented here.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol*h/ L
Arm/Group | BI 730357 + Itraconazole (T) | BI 730357 (R)
Number analyzed (Participants) | 14 | 14
nmol*h/ L | 64934.55 (NA) — Standard Error is Geometric standard error (gSE) = 1.10 | 6971.67 (NA) — Standard Error is Geometric standard error (gSE) = 1.10
Statistical Analysis 1: Comparison: BI 730357 + Itraconazole (T) vs BI 730357 (R); [analysis description as in outcome 1, analysis 1]; Test type: Other; gMean ratio (%) (T/ R) = 931.41, 90% CI 2-sided [785.19 to 1104.85], Standard Error of Mean 25.9 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: BI 730357: From first administration of BI 730357, up to 168 hours. Itraconazole: From first administration of itraconazole until second administration of BI 730357, up to 73 hours. BI 730357+ Itraconazole: From second administration of BI 730357 until 216 hours after the last administration of itraconazole, up to 18 days.
Description: Treated set (TS): The TS included all subjects who received at least 1 dose of trial medication.
Groups:
- Itraconazole: Participants were administered Itraconazole oral solution once daily on Day -3 to Day 1 before administration of 50 mg BI 730357 and on Day 2 to 9 after administration of BI 730357 in treatment period 2 only (T).
Arm/Group | BI 730357 (R) | Itraconazole | BI 730357 + Itraconazole (T)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 5/14 | 8/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 730357 (R) (N=14) | Itraconazole (N=14) | BI 730357 + Itraconazole (T) (N=14)
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 3
Presyncope (Nervous system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03782987/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT03782987/SAP_001.pdf